CLINICAL TRIAL: NCT05529654
Title: IMpella-Protected cArdiaC Surgery Trial (IMPACT)
Acronym: IMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VV-TMF-20447
Record Dates: First submitted 2022-08-24; First posted 2022-09-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Left Ventricular Dysfunction
Keywords: High-risk Cardiac Surgery; Low pre-operative left ventricular ejection fraction; Cardiopulmonary bypass (CPB); Temporary Mechanical Circulatory System (MCS)
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Impella Arm (Experimental): Impella 5.5 with SmartAssist
  Interventions: Device: Impella 5.5 with SmartAssist

INTERVENTIONS:
Device: Impella 5.5 with SmartAssist — For subjects enrolled in the Trial, the Impella 5.5 will be placed intra-operatively during the index cardiac surgical procedure

SUMMARY:
The purpose of this Trial is to demonstrate the safety and effectiveness of the use of Impella 5.5 in high-risk cardiac surgery patients, with the overall aim to evaluate if using Impella 5.5 with SmartAssist (Impella 5.5) peri-operatively improves early hemodynamics, end-organ function and clinical outcomes in patients with severely reduced LV function undergoing cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective single-armed Trial to demonstrate the safety and effectiveness of the use of Impella 5.5 in high-risk cardiac surgery patients. A concurrent Registry will also be performed to collect information on patients meeting Exclusion Criteria and those not approached for enrollment. The overall aim is to evaluate if using Impella 5.5 peri-operatively improves early hemodynamics, end-organ function and subsequent clinical outcomes in patients with severely reduced LV function undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamically stable patients undergoing one of the following cardiac surgery procedures on CPB including aortic cross-clamping and cardioplegic arrest:

   * Isolated CABG
   * Isolated mitral valve repair or mitral valve replacement (MVR)
   * Isolated biological aortic valve replacement (AVR)
   * At least two of the following: CABG, MVR, AVR, or tricuspid valve repair or replacement (TVR)
   * Additional concomitant procedures permitted:

     1. Atrial septal defect (ASD) or patent foramen ovale (PFO) repair or closure
     2. Atrial fibrillation ablation procedures
     3. Left atrial ablation (all forms including complete left/right side Cox Maze)
     4. Coronary endarterectomy
2. LVEF within 30 days before surgery of either:

   * ≤25% measured by echocardiogram or cardiac MRI, OR
   * LVEF ≤35%, measured as above, for patients with significant mitral regurgitation (MR 3+ or 4+) and planned corrective mitral valve surgery (including MV replacement or repair)

     * Any subject with EF <20% must have viability assessment performed to assess CABG candidacy (MRI preferred)
3. Age 18 years or older
4. Subject (or subject's LAR, if allowed by IRB) has signed Informed Consent Form

Exclusion Criteria:

1. Salvage operation (cardiac arrest within 24 hours prior to index surgery)
2. Unresponsive state within 24 hours of the time of surgery
3. Any inotrope within 72 hours of surgery
4. Any MCS device (such as IABP, ECMO, Impella®, CentriMag™ or TandemHeart®) in place at time of informed consent and less than 24 hours prior to index study procedure
5. RV dysfunction requiring mechanical or inotropic support pre-operatively and/or likely to be needed post-operatively
6. Index procedures requiring total circulatory arrest (TCA), such as aortic arch replacement, planned durable LVAD, durable RVAD, planned right-sided temporary mechanical support of any kind, total artificial heart (TAH), cardiac transplantation, pericardiectomy, pulmonary thromboendarterectomy and septal myectomy
7. Restrictive or obstructive cardiomyopathy, constrictive pericarditis, restrictive pericarditis, pericardial tamponade or other conditions in which cardiac output is dependent on venous return
8. Ventricular septal defect (VSD)
9. Stroke within 30 days of the index cardiac surgical procedure
10. Prior mantle field chest irradiation
11. Prior solid organ or hematologic transplantation (heart, kidney, liver, lung, pancreas, bone marrow) or durable LVAD
12. History of chronic dialysis
13. Pre-existing liver dysfunction defined as: Child-Pugh Class B or C
14. Pre-existing pulmonary disease requiring home oxygen or "severe pulmonary disease" determined by enrolling Investigator
15. Systemic active infection or evidence of systemic bacterial, fungal or viral infection within 72 hours before surgery (blood culture positive with leukocytosis)
16. Confirmed COVID-19 infection within two weeks prior to operation
17. Suspected or known pregnancy
18. Participation in the active treatment or follow-up phase of another interventional clinical trial of an investigational drug or device which has not reached its primary endpoint
19. Known contraindication to heparin; History of bleeding diathesis or known coagulopathy or will refuse blood transfusions
20. Inability to perform aortic cross-clamp, such as due to porcelain aorta
21. Any contraindication or inability to place Impella 5.5 (per the IFU), including LV thrombus and/or presence of a mechanical aortic valve
22. Any organ condition, concomitant disease (e.g., psychiatric illness, current severe alcoholism or current drug abuse, cancer, hepatic or kidney disease), with life expectancy of ≤2 years or other abnormality that itself or the treatment of which could interfere with the conduct of the trial or that, in the opinion of the investigator and/or Sponsor's medical monitor, would pose an unacceptable risk to the patient in the trial.
23. Patient has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with trial procedures
24. Patient belongs to a vulnerable population [Vulnerable patient populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Composite of All-Cause Mortality | 90 days
Stroke (as defined by STS) | 90 days
New requirement for Renal Replacement Therapy (RRT) | 90 days
Rate of Post-Cardiotomy Cardiac Failure | Hospital discharge, usually within 30 days
  The rate of post-cardiotomy cardiac failure evaluated at hospital discharge.

SECONDARY OUTCOMES:
Number of attempts to wean from CPB | Intra-op, usually within 1 day
Duration of mechanical ventilation | ICU discharge, usually within 30 days
Duration and dosages of inotropes and vasopressors. Duration of mechanical circulatory support (Hours) | ICU Discharge, usually within 30 days
  measured in number of hours of dosage
Acute Kidney Injury | within 7 days or at ICU Discharge (usually within 30 days)
  a modified KDIGO Stages 2-3
Vasoactive-inotropic score (VIS) | ICU Discharge, usually within 30 days
Cardiovascular mortality | Hospital discharge, usually within 30 days
Major Hemolysis | Hospital Discharge, usually within 30 days
  defined by MCS-ARC
Major Vascular Complications | Hospital Discharge, usually within 30 days
  defined by MCS-ARC
Major Bleeding | Hospital Discharge, usually within 30 days
  defined by STS
Length of ICU Stay | ICU Discharge, usually within 30 days
Length of Hospital Stay | Hospital Discharge, usually within 30 days
Quality of Life (QoL) assessed by KCCQ | 90 Days Post-Op
Physical Activity | 90 Days Post-Op
  Measured by (Katz Activities of Daily Living (ADL) and Lawton Instrumental ADL (IADL)
Technical Success | Intra-op, usually within 1 day
  The successful use of the Impella 5.5 device will be assessed by the proportion of patients who undergo successful Impella implant, as well as the proportion of patients demonstrating successful wean off CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Goldstein, MD, Principal Investigator — Montefiore Medical Center; Edward Soltesz, MD, Principal Investigator — The Cleveland Clinic; Hermann Reichenspurner, MD, PhD, Principal Investigator — University Heart & Vascular Center Hamburg
Locations (20):
- United States (20):
  - Cardiology Associates Research Group, Jonesboro, Arkansas
  - Keck School of Medicine, Los Angeles, California
  - Tri-City Medical Center, San Diego, California
  - NCH Rooney Heart Institute, Naples, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Mass General Hospital, Boston, Massachusetts
  - Brigham & Women's, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation/Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Health, New York, New York
  - New York- Presbyterian Hospital/ Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Centennial Heart Cardiovascular, Nashville, Tennessee
  - University of Texas Austin Dell Medical School/Ascension Texas, Austin, Texas
  - Baylor Scott and White - Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No